CLINICAL TRIAL: NCT00157989
Title: Safety and Feasibility of Controlled Tidal Volume Resuscitation of Preterm Infants ≤ 28 Weeks' Gestation: A Randomized Controlled Pilot Study
Brief Title: Pilot Study to Assess Safety and Feasibility of Resuscitation of Preterm Infants With Controlled Volume of Air/Oxygen
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 04-0164-A
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Resuscitation
Keywords: Infant, Premature
MeSH Terms: conditions — Premature Birth

INTERVENTIONS:
Procedure: Controlled tidal volume resuscitation

SUMMARY:
QUESTION:

Is controlled tidal volume delivery during the resuscitation of preterm infants < 28 weeks' gestation safe and feasible?

BACKGROUND AND RATIONALE: Current resuscitation of preterm neonates follows the Neonatal Resuscitation Program (NRP) guidelines. During initial resuscitation, neonates are bagged with self/flow inflating bags to achieve adequate chest rise, heart rate > 100 per minute and a pink color. When positive pressure ventilation is delivered with a bag, tidal volume is not measured. It is likely that high tidal volume is delivered to the neonate in order to achieve a rapid response. The evidence from human and animal model studies suggests that the initiation of mechanical ventilation and volutrauma associated with continued ventilation, are associated with an increase in pro-inflammatory mediators in the lungs of the preterm infants which induce pulmonary injury. This may interfere with the signaling involved in alveolarization, leading to a decrease in alveolar formation or maldevelopment of the alveoli, and subsequent evolution to chronic lung disease (CLD) or bronchopulmonary dysplasia (BPD).

OBJECTIVE: To evaluate the safety and feasibility of controlling tidal volume delivery (and limiting manual ventilation), during the resuscitation of preterm infants < 28 weeks' gestation.

STUDY DESIGN AND SETTING: A randomized controlled pilot study of 40 preterm neonates at the Mount Sinai Hospital.

RESEARCH PLAN: All eligible parents at risk for preterm delivery at < 28 weeks' gestation will be approached. After obtaining written informed consent, infants will be randomized to standard resuscitation according to NRP guidelines (control group) or resuscitation using controlled tidal volume ventilation (5 ml/kg) (study group), if they require resuscitation. Crossover to the control group will be allowed if there is clinical deterioration or no clinical improvement after 3 minutes of intervention.

OUTCOMES:

1. Primary: Apgar scores at 5,10, 15 and 20 minutes and pH, pO2, and pCO2 levels within 1 hour of resuscitation and at 4 hours of life.
2. Secondary: Durations of mechanical ventilation, continuous positive airway pressure support, low flow oxygen/air requirement; respiratory status of infant at 28 days postnatal and 36 weeks' corrected gestational age. Incidences of air leak, intraventricular haemorrhage and all causes of mortality before discharge from NICU will be compared.

DETAILED DESCRIPTION:
Design Randomized controlled pilot study.

Setting: The study will be conducted at the Mount Sinai Hospital (MSH), Toronto which is a tertiary care teaching hospital in the Greater Toronto Area. Approximately 50-75 neonates <28 weeks' completed gestation are delivered at MSH per year. The institute has expertise in the resuscitation of such preterm infants. All deliveries of preterm infants are attended by an experienced respiratory therapist, a resuscitation nurse, a neonatology fellow and a pediatric resident.

Inclusion Criteria:

All neonates born at <28 completed weeks' gestation according to early ultrasonographic estimation or maternal account of last menstrual period.

Exclusion Criteria:

1. Antenatally diagnosed congenital cardio-respiratory anomalies
2. Infants with known chromosomal or genetic abnormalities
3. A prior knowledge of significant fetal distress (diagnosed on the basis of cardiographic monitoring and defined as fetal heart rate <100 beats per minute and/or loss of beat to beat variability, and/or biophysical profile of <4/8)

Recruitment: Attending staff neonatologists, respiratory therapists and nursing staff at the MSH will be informed of the study. Parents of potentially eligible neonates will be identified by daily enquiry in the case room and NICU, and approached by one of the investigators after the NICU team has consulted the parents regarding medical aspects of preterm birth. The details of the study will be explained to parent(s) and informed written consent will be obtained. Where one of the investigators is responsible for the immediate care of the newborn infant, another investigator will obtain informed consent. Recruitment will continue until 40 subjects have completed the study.

Randomization: After obtaining the consent from the parent(s), a previously sealed envelope will be opened to identify the group to which the subject is randomized.

Subjects will be randomized to two arms:

1. The control group will be resuscitated as per NRP guidelines.
2. The study group will follow NRP guidelines except that immediately after initial unresponsiveness to bag and mask ventilation for 30 seconds, the infants will be intubated and controlled TV breaths will be delivered at 5 ml/kg using volume guarantee ventilator (Babylog 8000, Drager Inc; Chantilly, US).

Procedure: All deliveries will be attended as per the current NICU protocol. After the delivery, the neonate will be transferred to a radiant warmer, dried, suctioned, and evaluated for respiratory effort, heart rate, and colour. Further management will follow according to the group of allocation.

Control Group: The neonates assigned to the control arm of the study will be resuscitated as per the current NRP algorithm.7,8 The neonate will be intubated, as recommended in the guidelines, if he/she is apneic or gasping or have a heart rate <100 per minute or centrally cyanosed after 30 seconds of intermittent positive pressure (IPPV) with a bag and mask and 100% oxygen.7,8 Manual IPPV via neonatal flow-inflating resuscitation bag will continue after intubation. Correct tube placement will be verified by clinical examination. The recommended algorithm for heart rate <60 per minute will be followed. Once the infant has been stabilized (oxygen saturation 86-92%, heart rate maintained at >100 per minute and pink colour), he/she will be weighed (the resuscitaire has in built scales to obtain the weight without disconnecting the infants from the respiratory support).

Surfactant (BLESTM, BLES Biochemicals Inc, London, Ontario, Canada) will be administered according to the current NICU protocol at MSH. This protocol recommends surfactant administration within 15 minutes of delivery to all infants <27 weeks' gestation and to infants >27 weeks' gestation if FiO2 requirements are >35% and mean airway pressure is >7 cm of H2O. Five ml/kg of surfactant will be instilled via the endotracheal tube into the lungs in three aliquots using a precut nasogastric tube attached to a syringe. Each aliquot will be delivered with the infant lying in one of three head positions - supine, left lateral and right lateral. Between the administration of each aliquot, the neonate will continue to receive manual IPPV. After the administration of surfactant, the neonate will be attached to a ventilator. If for any reason the administration of surfactant is delayed, the infant will be attached to ventilator whenever the attending doctor feels it appropriate. Subsequent administration of surfactant in this group will follow similar procedural framework as outlined above.

Study Group: In the first minute, neonates in the study group will be resuscitated as per the current NRP algorithm, that is 30 seconds of IPPV using bag and mask ventilation will be allowed. Intubation will proceed only for infants who are apneic, gasping, who have heart rate <100 per minute or centrally cyanosed after 30 seconds of intermittent positive pressure (IPPV) with a bag and mask and 100% oxygen. Similar to the control group, a neonatal flow-inflating resuscitation bag will be used to deliver IPPV before intubation. However immediately post-intubation, infants in the study group will be attached to a ventilator kept ready with the following preset parameters: PEEP of 4 cmH2O, peak inspiratory pressure limit of 25 cm H2O, FiO2 at 100%, rate of 40 breaths per minute, flow rate of 5-10 L/min and inspiratory time of 0.35 seconds. An assist control volume guarantee mode will be used during the resuscitation. A volume guarantee ventilator (Babylog 8000, Drager Inc; Chantilly, US) will be used for the purpose of the study. The TV will be set at 5 ml/kg. An estimated weight will be used initially (according to either a recent estimated fetal weight on prenatal ultrasonogram or mean birth weight for the gestational weight [if the infant is assumed to be not growth restricted] or an estimate according to the attending team). Correct tube placement will be verified by clinical examination. The recommended algorithm for heart rate <60 per minute will be followed.

If an infant is not achieving TV of 5 ml/kg despite reaching upper pressure limit, visual assessment of chest wall movement will be carried out. If the chest expansion is inadequate, upper pressure limit will be increased by 5 cm of H2O. If the chest expansion is adequate, assessment of leakage of volume between inspiration and expiration will be checked on the display of the ventilator. If the leak is found to be >30%, the infant will be excluded from the study as he/she would be deemed unfit for the volume controlled ventilation. An adequate response will be considered when oxygen saturation is between 86-92%, heart rate maintained >100 per minute and pink color. Once the infant has been stabilized, he/she will be weighed using similar technique described in the control group without disconnecting from ventilator. At this time, the TV will be adjusted to reflect correct weight of the infant.

Similar criteria for the administration of surfactant in the control group will be applied to the study group. However, in order to avoid disconnection from the ventilator and administration of manual breaths, a closed suctioning adapter with an administration port (NeolinkTM Viasys MedSystems, Whoellng, IL, US) will be attached to the endotracheal tube. Five ml/kg of surfactant (BLESTM, BLES Biochemicals Inc, London, Ontario, Canada) will be delivered to the lungs in similar way while continuing mechanical ventilation at the same settings.

Procedures common to both groups: An oxygen saturation monitor, cardiac leads and end tidal CO2 leads will be attached to all infants at the earliest possible time. Continuous cardio-respiratory monitoring will ensue and at the end of the resuscitation period the data will be printed out. A naso/orogastric tube will be inserted. Umbilical arterial and umbilical venous catheters will be inserted as per the routine of the NICU. A chest X-ray will be done to assess endotracheal tube and catheter placement. Once stable, infants will be transferred to the NICU. Further respiratory management of all infants will be performed as deemed appropriate by NICU team and will be similar. (All infants are routinely ventilated with an aim to achieve 4-6 ml/kg of TV). Furthermore, all infants will receive head ultrasounds according to the current NICU practice.

Crossover: Crossover to the control group will be allowed 3 minutes after the onset of the intervention

1. If oxygen saturations increase by less than 20% (for starting values of <65%) or
2. If oxygen saturations are <80% (for starting values of >65%) or
3. If the heart rate <100 beats per minute or
4. If there is persistent central cyanosis in spite of resuscitation with 100% oxygen. In that event, the infant will be deemed a non-responder and manual ventilation will be allowed. However, the infant would be analyzed in the group of randomization (intention to treat analysis). The transition period to achieve normoxia and normocapnia may be longer in the study group patients. Therefore, patients in the intervention group may have slow but sustained improvement and would not be considered non-responders.

SAFETY: It is anticipated that there will be concerns that neonates in the study arm are not responding to resuscitation as rapidly as the neonates in the control arm of the study. By ensuring that the oxygen saturations are increasing, it is likely that we will avoid hypoxia. Mild hypercapnia, defined as a PaCO2 45-55 mmHg, provided the arterial pH is >7.25 is currently practiced in most NICUs and the evidence suggests no adverse effects. Continuous monitoring of leak will ensure that the lungs are not over distended.

A safety monitoring committee comprised of two neonatologists and a respiratory therapist not involved in the study will be convened to observe adverse events and provide recommendations about the study to the investigators. They will also report any concerns about the study to the Research Ethics Board. The clinical data for each infant requiring crossover to the control arm will be presented to the safety committee. The safety committee after reviewing the data will provide comments to the investigators as to whether the study should continue or not. The safety committee will be authorized to stop the study if it finds that the standard care of the infants in the study group is being jeopardized.

STATISTICAL ANALYSIS: Data will be analyzed using the statistical package SPSS (version 10, Chicago, IL, USA). Chi-square test for categorical variables and Student's t test for continuous variables will be used to compare the demographic characteristics in both groups. Intention to treat analysis will be performed; that is subjects will be analyzed in the same group of allocation even if they needed to cross over to control arm. Duration profiles of ventilatory requirement, CPAP requirement, and oxygen/air requirement in two groups will be compared using Student's t test. The number of subjects requiring switch over to the control group due to failure will be recorded. A priori analysis is also planned to compare the Apgar scores and first blood gas parameters after assessing the distribution and applying appropriate statistical transformation. A p value of < 0.05 will be considered significant for all analysis.

ELIGIBILITY:
Inclusion Criteria:

* All neonates born at <28 completed weeks' gestation according to early ultrasonographic estimation or maternal account of last menstrual period.

Exclusion Criteria:

* Antenatally diagnosed congenital cardio-respiratory anomalies
* Infants with known chromosomal or genetic abnormalities
* A prior knowledge of significant fetal distress (diagnosed on the basis of cardiographic monitoring and defined as fetal heart rate <100 beats per minute and/or loss of beat to beat variability, and/or biophysical profile of <4/8)

Ages: 0 Years to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 2004-10; Study Completion 2006-08

PRIMARY OUTCOMES:
Apgar scores at 5,10, 15 and 20 minutes and pH, pO2, and pCO2 levels within 1 hour of resuscitation and at 4 hours of life.

SECONDARY OUTCOMES:
Durations of mechanical ventilation, continuous positive airway pressure support, low flow oxygen/air requirement; respiratory status of infant at 28 days postnatal and 36 weeks' corrected gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Davey, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada